CLINICAL TRIAL: NCT06912919
Title: Effects of Low-intensity Blood Flow Restriction Exercise on Aerobic Capacity, Muscle Strength, Muscle Size, Biochemical-hormonal Parameters and Antioxidant Parameters in Overweight and Obese Individuals.
Acronym: YT BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul University Research Fund (Unknown)
Responsible Party: Principal Investigator, Yasin Atay, Medical Doctor, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: YT-1
Record Dates: First submitted 2025-03-13; First posted 2025-04-06 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-01

CONDITIONS: Obese Patients; Overweight (BMI > 25)
Keywords: Obesity; Blood Flow Restriction; Low Intensity Exercise; Antioxidant; Muscle Power; Cross Sectional Area; Hormone Profile; Overweight
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction (BFR) Aerobic Exercise Group (Experimental): 6 weeks, 3 days a week, 20 minutes of cycling exercise using 160-180 mmHg BFR.
  Interventions: Other: BFR-Aerobic Training
- Control Group (No BFR) (Experimental): 6 weeks, 3 days a week, 20 minutes of cycling exercise, no BFR.
  Interventions: Other: Aerobic Training Without BFR

INTERVENTIONS:
Other: BFR-Aerobic Training — Low-intensity cycling exercise with BFR (pressure of 160-180 mmHg) for 20 minutes, 3 days a week for 6 weeks.
  Arms: Blood Flow Restriction (BFR) Aerobic Exercise Group
Other: Aerobic Training Without BFR — Low-intensity cycling exercise (without BFR) for 20 minutes, 3 days a week for 6 weeks.
  Arms: Control Group (No BFR)

SUMMARY:
Participants will be selected from sedentary men aged 18-30 and over with a body mass index of 25. First, an informed consent form will be signed by the individuals. The 'International Physical Activity Questionnaire' will be applied to the participants and it will be ensured that the participants have not participated in vigorous and moderate activities and therefore are inactive or minimally active individuals. The study will consist of an intervention group and a control group, and the groups will be randomized via computer. The exclusion criteria of the study are that the participants do not have any known cardiac or pulmonary pathology and do not have any musculoskeletal disorders that will affect their participation in exercise. First, blood samples will be taken from the participants. They will be sent to the laboratory for examination of biochemical, hormonal and antioxidant parameters. Then, the muscle cross-sectional area and muscle thickness values of the rectus femoris muscle will be calculated from the participants with ultrasound measurements. After these procedures are completed, Vo2Max calculation will be performed on the participants with a cardiopulmonary exercise test. In addition, 40% of the Vo2Max value calculated in this test will be calculated and the pulse range to be used in the exercise will be determined. In the final stage, participants' strength isokinetic test and knee flexion extension strength and endurance values will be calculated.

After the evaluations are completed, individuals will start a 6-week exercise program. The intervention group will exercise with the blood flow restriction method under 160 mmHg pressure for the first 3 weeks and 180 mmHg pressure for the last 3 weeks. The device will be applied by placing it at the most proximal point of the thigh. The control group will do the same exercise without restricting blood flow. Both groups will be followed for 6 weeks with a 5-minute warm-up followed by a 20-minute exercise program. Participants will report their fatigue with the Borg scale after each exercise session.

After the exercise sessions are completed, blood will be taken on an empty stomach within 24 hours of the last exercise. Then, muscle size measurement with ultrasound, Vo2Max calculation and isokinetic test power calculation will be noted, respectively. The values obtained will be compared with the initial values.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-30 Gender: Male Body Mass Index (BMI) ≥ 25 kg/m² Inactive or minimally active individuals (assessed with the International Physical Activity Questionnaire - IPAQ) No history of metabolic, cardiovascular or neuromuscular disease Not taking any medication that affects metabolism, hormones or muscle function Able to participate in a 6-week exercise program

Exclusion Criteria:

Having a cardiac or respiratory complaint Having a known chronic disease Having a medication used regularly

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — For study symmetry, only male sedentary overweight and obese individuals were selected.
Enrollment: 34 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Change in VO2Max | 6 weeks (pre-post test)
  VO2Max (ml/kg/min) will be measured by indirect gas analysis and compared before and after exercise.
Change in Isokinetic Muscle Strength | 6 weeks (pre-post test)
  Quadriceps and hamstring strength will be evaluated with an isokinetic dynamometer.
Change in Muscle Cross-Sectional Area (CSA) | 6 weeks (pre-post test)
  The muscle cross-sectional area (cm²) of the Rectus Femoris will be measured by ultrasound (USG) and its change will be evaluated.
Change in Muscle Thickness (MT) | 6 weeks (pre-post test)
  The muscle thickness (mm) of the Rectus Femoris will be measured by ultrasound (USG) and its change will be evaluated.

SECONDARY OUTCOMES:
Change in Oxidative Stress and Antioxidant Capacity | 6 weeks
  Systemic oxidative stress and total antioxidant capacity will be assessed through blood biomarkers before and after the intervention.
Change in Cortisol Levels | 6 weeks
  Cortisol levels will be measured with a pre- and post-exercise blood test.
Change in Glucose Levels | 6 weeks
  Glucose levels will be measured with a pre- and post-exercise blood test.
Change in Creatine Kinase Levels | 6 weeks
  Creatine kinase levels will be measured with a pre- and post-exercise blood test.
Change in Cholesterol Levels | 6 weeks
  Cholesterol levels will be measured with a pre- and post-exercise blood test.
Change in Triglyceride Levels | 6 weeks
  Triglyceride levels will be measured with a pre- and post-exercise blood test.
Change in Testosterone Levels | 6 weeks
  Blood samples will be collected to measure testosterone levels before and after the intervention.
Change in Luteinizing Hormone (LH) Levels | 6 weeks
  Luteinizing hormone (LH) levels will be measured with a pre- and post-exercise blood test.
Change in Follicle-Stimulating Hormone (FSH) Levels | 6 weeks
  Follicle-stimulating hormone (FSH) levels will be measured with a pre- and post-exercise blood test.
Change in Dehydroepiandrosterone Sulphate (DHEAS) Levels | 6 weeks
  Dehydroepiandrosterone sulphate (DHEAS) levels will be measured with a pre- and post-exercise blood test.
Change in Sex Hormone-Binding Globulin (SHBG) Levels | 6 weeks
  Sex hormone-binding globulin (SHBG) levels will be measured with a pre- and post-exercise blood test.
Change in Free Androgen Index (FAI) Levels | 6 weeks
  Free androgen index (FAI) levels will be measured with a pre- and post-exercise blood test.
Change in BMI (kg/m²) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Faculty of Medicine. Sports Medicine Department, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murakami K, Okimoto T, Kodama M, Tanahashi J, Yasaka S, Inoue K, Uchida M, Anan J, Mizukami K, Abe T, Watada M, Fujioka T. Helicobacter pylori and NSAID-induced gastric ulcer in a Japanese population. J Gastroenterol. 2009;44 Suppl 19:40-3. doi: 10.1007/s00535-008-2259-5. Epub 2009 Jan 16. PMID 19148792
- [Background] Kim D, Singh H, Loenneke JP, Thiebaud RS, Fahs CA, Rossow LM, Young K, Seo DI, Bemben DA, Bemben MG. Comparative Effects of Vigorous-Intensity and Low-Intensity Blood Flow Restricted Cycle Training and Detraining on Muscle Mass, Strength, and Aerobic Capacity. J Strength Cond Res. 2016 May;30(5):1453-61. doi: 10.1519/JSC.0000000000001218. PMID 26439780